CLINICAL TRIAL: NCT03719885
Title: Prospective Controlled Study of Intranasal Tear Neurostimulation for Sjogrens Patients With Dry Eye Disease
Brief Title: TrueTear in Sjogren's Disease Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Pennsylvania (Other)
Collaborators: Allergan (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 830076
Record Dates: First submitted 2018-10-19; First posted 2018-10-25 (Actual); Results first posted 2020-08-25 (Actual); Last update posted 2023-07-07 (Actual); Status verified 2023-07

CONDITIONS: Dry Eye Syndromes; Sjogren's Syndrome
MeSH Terms: conditions — Dry Eye Syndromes; Sjogren's Syndrome

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (1):
- Intervention (Experimental)
  Interventions: Device: TrueTear Intranasal Tear Neurostimulator

INTERVENTIONS:
Device: TrueTear Intranasal Tear Neurostimulator — This study will evaluate the immediate tear production resulting from use of intranasal tear neurostimulation in patients with Sjogren's disease

SUMMARY:
The purpose of this study is to evaluate acute tear production produced by the intranasal tear neurostimulator in participants with Sjögrens syndrome and aqueous tear deficiency. Our primary goal is to evaluate whether Sjögrens patients respond to this intervention and whether there is a baseline tear production level below which these patients do not respond.

ELIGIBILITY:
Inclusion Criteria:

* Subjects with Sjögren's syndrome based on American-European Consensus Group (AECG) American College of Rheumatology (ACR), or American College of Rheumatology/European League Against Rheumatism (ACR/EULAR) criteria
* Baseline Schirmer score (with topical anesthesia) of ≤10 mm/5 min and retest value (during nasal stimulation with cotton swab) of at least 4 mm/5min higher than baseline value
* Baseline Ocular Surface Disease Index® (OSDI) total score ≥13
* Age greater than or equal to 22 years old
* Able to complete questionnaires independently
* Willing to sign the informed consent and deemed capable of complying with the requirements of the study protocol

Exclusion Criteria:

* Use of any topical ophthalmic medication, including artificial tears, within 4 hours of either visit
* Chronic or recurrent epistaxis, coagulation disorders or other conditions that, in the opinion of the investigator, may lead to clinically significant increased bleeding
* Use of systemic anticoagulants
* Nasal or sinus surgery including nasal cautery or significant trauma
* Severely deviated septum
* Cardiac demand pacemaker, implanted defibrillator or other implanted electronic device
* Have an active implanted metallic or active implanted electronic device in the head, a cardiac demand pacemaker, or an implanted defibrillator
* Known hypersensitivity to any of the procedural agents or materials in the study device that contact the nasal mucosa
* Corneal transplant in either or both eyes
* Participation in any clinical trial within 30 days of the Screening Visit
* A woman who is pregnant, planning a pregnancy, or nursing at the Screening Visit

Min Age: 22 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 55 (Actual)
Dates: Start 2018-12-01 (Actual); Primary Completion 2019-04-25 (Actual); Study Completion 2019-12-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Giacomina Massaro-Giordano, MD, Principal Investigator — Scheie Eye Insitute, University of Pennsylvania
Locations (1):
- Scheie Eye Institute, University of Pennsylvania, Philadelphia, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Study Group: The participants recruited for this study were those who were 22 years or older, had a clinical diagnosis of Sjogren's Syndrome (SS), and produced 10 mm. or less of tears over the course of 5 minutes (measured using Schirmer strips). They also had to have an OSDI score ≥13.
Period: Overall Study
Arm/Group | Study Group
Started | 55
Completed | 35
Not Completed | 20

BASELINE CHARACTERISTICS:
Population: Same as assignment in Participant Flow
Groups:
- Study Group: The participants recruited for this study were those who had a clinical diagnosis of Sjogren's Syndrome (SS) and produced 10 mm. or less of tears over the course of 5 minutes (measured using Schirmer strips).
Arm/Group | Study Group
Number analyzed (Participants) | 35
Age, Continuous [Mean (Standard Deviation); unit: years] | 57.1 (11.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 35
  Male | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1
  Not Hispanic or Latino | 33
  Unknown or Not Reported | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 2
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 5
  White | 26
  More than one race | 1
  Unknown or Not Reported | 1
Year of Sjogren's diagnosis [Count of Participants; unit: Participants]
  Prior to 2000 | 3
  2000 - 2010 | 11
  After 2010 | 21
OSDI Score [Mean (Standard Deviation); unit: units on a scale] — [low of 0, high of 100] Higher score means more affected by dry eye symptoms, lower score means less affected by dry eye symptoms- OSDI score defined the ocular surface as normal (0-12 points) or as having mild (13-22 points), moderate (23-32 points), or severe (33-100 points) disease.
  units on a scale | 50.5 (21)

OUTCOME MEASURES:

1. Primary Outcome: Schirmer Testing
Description: Tear production measured immediately following intranasal tear neurostimulation. For this measurement, Schirmer strips (small strips of paper with measurements on them) are placed in the corner of each eye. The amount of wetting of the Schirmer strips is measured in millimeters. Wetting of less than 5 mm is indicative of deficient tear production.
Time Frame: Immediately following the procedure (ie immediately following use of the device)
Measure: Mean (Standard Deviation); unit: mm.
Groups:
- Intervention: TrueTear Intranasal Tear Neurostimulator: This study will evaluate the difference between active and control applications in tear production during active stimulation as measured by Schirmer testing
Arm/Group | Intervention
Number analyzed (Participants) | 35
mm.
  Cotton Swab | 10.2 (1.3)
  Extranasal Application | 0.8 (0.8)
  Intranasal Application | 13.5 (1.6)

2. Secondary Outcome: Clinically Significant Changes in Visual Acuity
Description: Clinically significant change in Best corrected visual acuity (BCVA)- this measurement was taken to determine if a significant change in BCVA was noted for participants. If a clinically significant change was noted (greater or equal to 2 lines of vision) then a subject would be listed in the data table below.
Time Frame: Immediately following the procedure (ie immediately following use of the device)
Population: Participants' eyes were examined pre and post active application to confirm that the device did not cause any changes to the participant's vision. A serious change in vision would have been reported as an adverse event
Measure: Count of Participants; unit: Participants
Arm/Group | Intervention
Number analyzed (Participants) | 35
Participants | 0

3. Secondary Outcome: Clinically Significant Changes in Slit Lamp Exam
Description: Clinically significant changes in slit lamp examination . Subjects who experienced clinically significant changes would be represented in the data table below.
Time Frame: Immediately following the procedure (ie immediately following use of the device)
Population: Eyes were examined pre and post active application to confirm that the device did not cause any changes to the physical structure or appearance of the eyes
Measure: Count of Participants; unit: Participants
Groups:
- Intervetion: TrueTear Intranasal Tear Neurostimulator: This study will evaluate the immediate tear production resulting from use of intranasal tear neurostimulation in patients with Sjogren's disease
Arm/Group | Intervetion
Number analyzed (Participants) | 35
Participants | 0

4. Secondary Outcome: Number of Adverse Events
Description: Pain, headache, nosebleed, etc felt to be associated with use of the device
Time Frame: Immediately following the procedure (ie immediately following use of the device)
Population: All participants who used the device were observed for any adverse events
Measure: Number; unit: occurance of adverse event
Arm/Group | Intervention
Number analyzed (Participants) | 35
occurance of adverse event | 1

ADVERSE EVENTS:
Time Frame: Adverse events were collected throughout the duration of the study (from the time the patient was enrolled in the study until they completed visit 2). We also provided patients with our contact information, in case they experienced any adverse events in the days following visit 2.
Description: The adverse event data was collected immediately following the event. The subject was also called a week later to ensure that the issue had resolved.
Arm/Group | Study Group
All-Cause Mortality (participants affected / at risk) | 0/55
Serious Adverse Events (participants affected / at risk) | 0/55
Other Adverse Events (participants affected / at risk) | 1/55
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Study Group (N=55)
Small conjunctival hemorrhage (Eye disorders) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2019-09-10): https://cdn.clinicaltrials.gov/large-docs/85/NCT03719885/Prot_SAP_000.pdf
  • Informed Consent Form (2018-11-19): https://cdn.clinicaltrials.gov/large-docs/85/NCT03719885/ICF_001.pdf